CLINICAL TRIAL: NCT05815511
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Effect of a Probiotic Mixture on the Evolution and Treatment of Rosacea
Brief Title: Clinical Trial to Evaluate the Effect of a Probiotic Mixture on the Rosacea Evolution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionou Research, S.L. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROS.PROB
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Rosacea; Rosacea Papular Type; Rosacea, Papulopustular
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Intervention Model Description: Clinical trial randomized, double-blind, and placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic group (Experimental): Probiotic mixture in oral capsule format with selected strains in concentrations equal to or greater than 1x10^10 cfu/dose.
  Interventions: Dietary Supplement: Probiotic mixture
- Placebo group (Placebo Comparator): Maltodextrin in oral capsule format
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic mixture — Oral capsule consumption once a day for 12 weeks
  Arms: Probiotic group
Dietary Supplement: Placebo — Oral capsule consumption once a day for 12 weeks
  Arms: Placebo group

SUMMARY:
The clinical trial has a randomized, double-blind, placebo-controlled design, in which the aim is to evaluate the effect of a probiotic mix, with a 12-week treatment, on the evolution of rosacea.

This 12 weeks of treatment are structured into three visits: Visit 1 (initial; week 0), Visit 2 (intermediate; week 6) and Visit 3 (final; week 12).

DETAILED DESCRIPTION:
The three visits that make up the study and the actions to be carried out in each of them are described below:

Visit 1 (initial; week 0)

Once the informed consent is signed, a doctor trained for the study performs the initial interview where it is verified that the patient meets all the inclusion criteria and none of the exclusion criteria and their medical history.The investigator will proceed to assign the patient the next study participant number and, according to a previously prepared randomization list, the treatment that they will receive during the study will be assigned.

The investigator will assess the severity and symptoms of rosacea according to the Investigator's Global Assessment (IGA) and Clinician Erythema Assessment (CEA) scales. The patient will also complete a questionnaire to assess the impact on quality of life due to the disease: Dermatology Life Quality Index (DLQI).

Visit 2 (intermediate; week 6)

In this intermediate visit, in addition to assessing the symptoms of the disease with the detailed scales, the investigator will record the adverse events reported by the patient, as well as the concomitant treatments used.

Also, the treatment compliance rate will be calculated by counting the capsules returned by the patient.

Visit 3 (final; week 12)

In the final visit, the same actions will be carried out as in the intermediate visit, evaluating the severity of the disease and the remaining capsules will be collected, to calculate treatment compliance, concomitant treatments and adverse events.

Visit 4 (post-treatment follow-up; week 24)

During this visit, the symptoms of the disease will be assessed with the two scales used in the study and the treatments that the patient has required during the 12 weeks after the end of the study treatment will be counted.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes of an age equal to or greater than 18 years.
* Patients diagnosed with papulopustular rosacea with a minimum score of 2 points according to the Investigator's Global Assessment (IGA) index.
* Signature of informed consent by the patient

Exclusion Criteria:

* Pregnant, lactating, and/or women who do not agree to use an effective contraceptive method during the development of the study.
* Allergy and/or intolerance to any of the components of the product under study.
* Consumption of antibiotics in the previous two weeks.
* Consumption of probiotics in the previous two months.
* Isotretinoin use in the previous six months.
* Light procedures (IPL, laser, Kleresca) in the previous three months.
* Participation in other clinical studies in the previous two months.
* Other dermatological pathologies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Number and percentage of cases responding to the treatment according to the Investigator's Global Assessment (IGA) index score, comparing the baseline with the visits at 6 and 12 weeks | 12 weeks
  IGA index measures the severity of rosacea
  Score range is from 0 to 6 according to the severity of the disease
  0=clear; 1=minimum; 2=mild; 3=mild-moderate; 4=moderate; 5=moderate-severe; 6=severe
  It will be considered a treatment response in IGA scale when the participant improves by at least 2 categories in this index and the final score is 0-1 points (clear and almost clear)

SECONDARY OUTCOMES:
Number and percentage of cases responding to the treatment according to the IGA index score, analyzing the cases that received any topical or systemic treatment, comparing the baseline with the visits at 6 and 12 weeks | 12 weeks
  The treatments considered will be any topical or systemic treatment
Number and percentage of cases responding to the treatment according to the IGA index score, analyzing the cases that received systemic treatment, comparing the baseline with the visits at 6 and 12 weeks | 12 weeks
  The treatments considered will be any systemic treatment
Number and percentage of cases that need any treatment (topical or systemic) and number of days during the treatment period (12 weeks) | 12 weeks
  The number of treatment days and the number of participants prescribed treatment by the dermatologist will be counted
  The treatments considered will be any topical or systemic treatment
Number and percentage of cases that need systemic treatment and number of days during the treatment period (12 weeks) | 12 weeks
  The number of treatment days and the number of participants prescribed systemic treatment by the dermatologist will be counted
  The treatments considered will be any systemic treatment
Number and percentage of cases that need topical treatment and number of days during the treatment period (12 weeks) | 12 weeks
  The number of days and the number of participants prescribed topical treatment by the dermatologist will be counted
  The treatments considered will be any topical treatment
Number and percentage of cases responding to the treatment according to the Dermatology Life Quality Index (DLQI) at 6 and 12 weeks | 12 weeks
  DLQI measures the impact rosacea has on your quality of life
  The index has 10 questions. Each question answered with "Very much" is counted with 3 points, "A lot" with 2, "Little" with 1, and "Not at all" as 0.
  The score obtained can range between 0 and 30 points, this being the worst possible score.
  It will be considered a treatment response in DLQI scale when the score is 0-5 points (no effect or mild effect in the quality of life)
Number and percentage of cases responding to the treatment according to the IGA index score, comparing the baseline with the visit at 24 weeks (post-treatment follow-up) | 24 weeks
  IGA index measures the severity of rosacea
  Score range is from 0 to 6 according to the severity of the disease
  0=clear; 1=minimum; 2=mild; 3=mild-moderate; 4=moderate; 5=moderate-severe; 6=severe
  It will be considered a treatment response when the participant improves by at least 2 categories in this index and the final score is 0-1 points (clear and almost clear)
Number and percentage of cases requiring any treatment (topical or systemic), along with the number of days, covering the total period (24 weeks) and the post-treatment follow-up period (from week 12 to 24) | 24 weeks
  The number of treatment days and the number of participants prescribed treatment by the dermatologist will be counted
  The treatments considered will be any topical or systemic treatment
Number and percentage of cases requiring systemic treatment, along with the number of days, covering the total period (24 weeks) and the post-treatment follow-up period (from week 12 to 24) | 24 weeks
  The number of treatment days and the number of participants prescribed systemic treatment by the dermatologist will be counted
  The treatments considered will be any systemic treatment
Number and percentage of cases requiring topical treatment, along with the number of days, covering the total period (24 weeks) and the post-treatment follow-up period (from week 12 to 24) | 24 weeks
  The number of treatment days and the number of participants prescribed topical treatment by the dermatologist will be counted
  The treatments considered will be any topical treatment
Study treatment compliance rate at 6 and 12 weeks. | 12 weeks
  The treatment adherence is collected, checking the number of remaining capsules in each of the visits

OTHER OUTCOMES:
Number of adverse events at 6 and 12 weeks | 12 weeks
  Adverse events reported by patients during follow-up at week 6 and week 12 visits are recorded

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Eguren Dermatology and Aesthetics Clinic, Madrid, Madrid
  - MiBioPath UCAM Research Group, Murcia, Murcia
  - Gavín Dermatologists Clinic, Vigo, Pontevedra